CLINICAL TRIAL: NCT00934401
Title: Positron Emission Mammography With 3'-Deoxy-3'-[18F] Fluorothymidine (FLT PEM) for Evaluation of Response to Neoadjuvant Chemotherapy in Breast Cancer
Brief Title: Positron Emission Mammography With Fluorothymidine (FLT) to Evaluate Treatment Response to Chemotherapy in Breast Cancer
Status: Withdrawn | Type: Observational
Why Stopped: poor accrual
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Yusuf Menda, Associate Professor, University of Iowa
Other Study IDs: 200903755
Record Dates: First submitted 2009-07-06; First posted 2009-07-08 (Estimated); Last update posted 2016-07-11 (Estimated); Status verified 2016-07

CONDITIONS: Breast Neoplasms
Keywords: FLT; fluorolabeled thymidine; breast cancer; Positron-Emission Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Positron Emission Tomography Imaging with 3-Deoxy-3'-[18F]Fluorothymidine (FLT) can selectively identify proliferating and non-proliferating tissues, including tumors. FLT uptake in the tumor is an indirect marker of DNA synthesis activity, which is a target of chemotherapy. Our hypothesis is that early change in FLT uptake in tumor with chemotherapy will predict pathological response to neoadjuvant therapy in breast cancer. Tumor uptake of FLT will be imaged and measured with positron emission mammography (PEM), a PET scanner optimized for breast imaging with a significantly improved resolution compared to conventional whole-body PET imaging systems.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and willingness to sign a written informed consent document.
2. Subject must have histologically confirmed breast cancer.
3. Subject must be scheduled to receive neoadjuvant chemotherapy followed by surgery for their standard cancer care. Treatment decisions will be made by the treating surgeon and the medical oncologist.
4. Females at least 18 years of age.
5. Karnofsky at least 60% at time of screening.
6. Life expectancy of greater than 6 months.
7. Subject must have normal organ and marrow function (as defined below) within 30 days of study enrollment:

   * leukocytes at least 3,000/microL
   * absolute neutrophil count at least 1,500/microL
   * platelets at least 100,000/microL
   * total bilirubin Equal or less than 1.0 mg/dl
   * AST(SGOT) no greater than 2.5 X institutional upper limit of normal
   * ALT (SGPT) no greater than 2.5 X institutional upper limit of normal
   * Creatinine Equal or less than 1.4 mg/dl
   * BUN Equal or less than 20 mg /dl
8. The effects of FLT on the developing human fetus are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately. A screening urine hCG will be administered in the Nuclear Medicine to women of childbearing potential before each FLT scan and pregnant women will not be accepted as subjects in this study.

Exclusion Criteria:

1. Subjects who have had chemotherapy or radiotherapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier.
2. Subject with a Karnofsky score of below 60.
3. Pregnant women are excluded from this study. FLT PET has potential for teratogenic effects. Because there are potentially unknown risks for adverse events in nursing infants secondary to treatment of the mother with FLT, breastfeeding should be discontinued if the mother is imaged with FLT and may not resume for 48 hours after the FLT imaging.
4. Subjects taking nucleoside analog medications such as those used as antiretroviral agents.

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women diagnosed with breast cancer whose recommended treatment is neoadjuvant chemotherapy followed by surgical resection.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2009-07; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Uptake of FLT (SUV) within the tumor | 20 mintues and 60 minutes post injection

SECONDARY OUTCOMES:
Pathologic tumor response | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf Menda, M.D., Principal Investigator — The University of Iowa Hospitals & Clinics
Locations (1):
- The University of Iowa Hospitals & Clinics PET Center, Iowa City, Iowa, United States